CLINICAL TRIAL: NCT00915239
Title: Symptom Evaluation After Cessation of a Proton Pump Inhibitor in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Einar Björnsson, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SUS/KUS2
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2009-06-05 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pantoprazole (Active Comparator)
  Interventions: Drug: Pantoprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pantoprazole — 40 mg pantoprazole once daily for 28 days
  Arms: Pantoprazole
Drug: Placebo — identical placebo once daily for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether proton pump inhibitor (PPI) induced hypersecretion leads to acid related symptoms after treatment in healthy volunteers.

DETAILED DESCRIPTION:
Treatment with proton pump inhibitors (PPI) has been shown to cause rebound hypersecretion of gastric acid. The clinical significance of this phenomenon is however unclear. This study aims to examine whether or not healthy volunteers, who over a relatively short period of time treated with a PPI, develop dyspeptic symptoms after cessation of therapy. Dyspeptic symptoms will be measured subjectively using a validated questionnaire, which is filled out each day. Gastric acid will be measured indirectly with measurement of acid secretion markers (Gastrin and chromogranin-A).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* 18-70 years of age
* Informed consent
* No prior history of any GI disorder

Exclusion Criteria:

* Dyspeptic complaints
* H. pylori infection
* Ongoing treatment with pain-relieving medications (i.e., NSAID)
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To evaluate whether healthy volunteers, treated with PPI for four weeks, develop acid-related symptoms after cessation of PPI therapy.

SECONDARY OUTCOMES:
To evaluate whether there is a correlation between markers for acid secretion such as gastrin and chromogranin-A and the development of dyspeptic symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Univeristy Hospital, Gothenburg, Gothenburg, Sweden